CLINICAL TRIAL: NCT07097181
Title: The Effect of Sensory Awareness Education on Female Students' Body Awareness and Premenstrual Symptom Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Associate Professor Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBU-AYDINKARTAL-014
Record Dates: First submitted 2024-12-08; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: for Girls; Sensory Awareness Training; Body Awareness; Premenstrual Syndrome; Effect
Keywords: sensory awareness; education; student; premenstrual syndrome
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: Sensory awareness training was given to the female students in the intervention group of the research for 4 weeks.
  training will be given. Training contents, Sensory System Training Presentation, Proprioception and Kinesthesia Sense Training Presentation, Interoception Sense Training Presentation will be held later.
  Graded Sensory Discrimination, Graded Motor Imagery (DMI), interoception consisting of awareness training, interoceptive awareness exercises and home exercises program.
  A protocol for training and body awareness training will be implemented.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (n:90) (No Intervention): No educational intervention will be made to the students in the control group.
- web-based sensory awareness training (n:90) (Experimental): Female students in the intervention group will receive sensory awareness training for four weeks. The training content will include presentations on the Sensory System, Proprioception and Kinesthesia, and Interoception. Following these presentations, a protocol focusing on body awareness will be implemented. This protocol will consist of graded sensory discrimination, graded motor imagery (GMI), interoception awareness training, interoceptive awareness exercises, and a home exercise program. Each training session will be planned to last 60 minutes.
  A pre-training briefing session will be held with female students who volunteer to participate and are assigned to the intervention group.
  Interventions: Behavioral: web-based sensory awareness training

INTERVENTIONS:
Behavioral: web-based sensory awareness training — The girl in the intervention group of the study 4 weeks to inform students, raise awareness and provide sensory education. Sensory awareness training will be provided throughout. Presentations to inform during training will be done, then Graded Sensory Discrimination, Graded Motor Imagery (DMI) and a home exercise program, as well as a body awareness training program.
  protocol will be applied.
  Arms: web-based sensory awareness training (n:90)

SUMMARY:
This research investigates the effects of web-based sensory awareness training on female students' body movements.

In order to examine its effect on awareness and premenstrual symptom levels. planned. H0a = Body awareness levels of female students who receive and do not receive sensory awareness training. There is no difference between.

H1a = Body awareness levels of female students who receive and do not receive sensory awareness training. There is a difference between .

H0b = Premenstrual symptoms of female students who received and did not receive sensory awareness training. There is no difference between the levels.

H1b = Premenstrual symptoms of female students who receive and do not receive sensory awareness training. There is a difference between the levels.

Participants will be given sensory awareness training for 4 weeks and female students will be given "Premenstrual Syndrome Scale" and "Very" before the training and 4 weeks after the first training.Dimensional Body Awareness Assessment-II Scale" will be applied

DETAILED DESCRIPTION:
The study will be conducted online via https://teams.microsoft.com/v2/. Female first-year students from the Midwifery Department and the Physiotherapy and Rehabilitation Department of SBÜ Hamidiye Faculty of Health Sciences who volunteer to participate will be assigned to the intervention group (n=90) and control group (n=90) using random numbers generated via https://www.randomizer.org/ by the researchers. All participants will complete an introductory information form.

Female students in the intervention group will receive sensory awareness training for four weeks. The training content will include presentations on the Sensory System, Proprioception and Kinesthesia, and Interoception. Following the presentations, a protocol focusing on body awareness will be implemented, including graded sensory discrimination, graded motor imagery (GMI), interoception awareness training, interoceptive awareness exercises, and home exercise programs. Each training session will be planned to last 60 minutes.

A pre-training briefing session will be held with the female students assigned to the intervention group who volunteer to participate. The "Premenstrual Syndrome Scale" and the "Multidimensional Assessment of Interoceptive Awareness-II Scale" will be administered to the students before the training and four weeks after the first session. Each training session will be conducted once a week and will be limited to 60 minutes. The study forms will be administered to participants in person.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research.
* University of Health Sciences, Hamidiye Faculty of Health Sciences, Department of Midwifery Being an active student in the first grade.
* University of Health Sciences, Hamidiye Faculty of Health Sciences, Physiotherapy and Being an active female student in the first year of the Department of Rehabilitation.
* Having internet access.
* Having a smart mobile phone.

Exclusion Criteria:

* University of Health Sciences, Hamidiye Faculty of Health Sciences, Department of Midwifery Being a passive student in the first grade.
* University of Health Sciences, Hamidiye Faculty of Health Sciences, Physiotherapy and Being a passive female student in the first year of the Rehabilitation Department.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 6 week
  In this form created by researchers based on the literature, It includes questions about the participants' age, high school they graduated from, menstrual period and symptoms.
  is taking.
Premenstrual Syndrome Scale (PMSS) | 6 week
  The scale was developed by Gençdoğan in 2006. It consists of 44 items and is designed in a five-point Likert format. The scoring of the scale is as follows: "Never" is scored as 1 point, "Rarely" as 2 points, "Sometimes" as 3 points, "Often" as 4 points, and "Always" as 5 points. The scale includes nine subdimensions:Fatigue ,Depressive Affect,Depressive Thoughts,Anxiety ,Irritability ,Appetite Changes ,Pain ,Sleep Changes ,Bloating.The PMS Scale (PMSÖ) score is obtained by summing the scores of these subdimensions. The scale is administered by asking the individual to respond based on their experience during the week before their menstruation. The total score ranges from a minimum of 44 to a maximum of 220. A higher score indicates more severe premenstrual symptoms.
Multidimensional Body Awareness Assessment-II Scale | 6 week
  Body Awareness has multiple developed by Mehling, Acree, Stewart, Silas and Jones to measure the dimensions of The Turkish adaptation of the scale was made by Mungurlar and Kahya. Scale, 37 It is a self-report scale consisting of one item and eight factors. These factors; "Noticing", "Attention "Not Distracting", "Not Worrying", "Regulating Attention", "Emotional Awareness", "Self-Regulation", "Listening to the Body" and "Trusting". Evaluation of the scale is 1-5 points and is made by averaging the scoring factors separately. of scale Validity reliability Cronbach's alpha coefficient was determined as 0.88. As the score obtained from the scale increases, it means that people have more positive body awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)